CLINICAL TRIAL: NCT06774222
Title: A Phase II, Single-Arm, Single-Center Study of Fruquintinib Combined With Standard Chemotherapy for Postoperative Treatment of HER2-Negative Gastric Cancer Patients With Poor Tumor Regression Grade.
Brief Title: A Study of Fruquintinib Plus Chemotherapy for Postoperative Treatment of HER2-Negative Gastric Cancer With Poor TRG
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-421
Record Dates: First submitted 2024-12-12; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-11

CONDITIONS: Gastric/Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — HMPL-013

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Fruquintinib Combined with Standard Chemotherapy
  Interventions: Drug: Fruquintinib

INTERVENTIONS:
Drug: Fruquintinib — Fruquinitinib: Take 4 mg QD for 2 weeks and stop for 1 week, every 3 weeks for a cycle; Standard chemotherapy: The selection of drugs is recommended by the 2024CSCO Guidelines for the Diagnosis and Treatment of Gastric Cancer, including SOX, XLOX or S-1, and the treatment cycle is one every 3 weeks
  Other Names: HMPL-013

SUMMARY:
Given that a significant proportion of locally advanced gastric cancer patients still die from tumor recurrence after surgery, with long-term therapeutic outcomes stagnating and difficult to further improve, especially for patients with poor tumor regression grade (TRG) after surgery, this study aims to explore a new model of adjuvant therapy by conducting research on the use of Fruquintinib in combination with standard chemotherapy for postoperative treatment of HER2-negative gastric cancer patients with poor TRG, in order to bring greater survival benefits to patients.

DETAILED DESCRIPTION:
Given that a significant proportion of locally advanced gastric cancer patients still die from tumor recurrence after surgery, with long-term therapeutic outcomes stagnating and difficult to further improve, especially for patients with poor tumor regression grade (TRG) after surgery, this study aims to explore a new model of adjuvant therapy by conducting research on the use of Fruquintinib in combination with standard chemotherapy for postoperative treatment of HER2-negative gastric cancer patients with poor TRG, in order to bring greater survival benefits to patients. The primary endpoint of this study is to evaluate the recurrence-free survival (RFS) in patients with poor TRG after neoadjuvant chemotherapy for gastric cancer who receive adjuvant therapy with Fruquintinib combined with standard chemotherapy postoperatively. Secondary endpoints include overall survival (OS) and safety .

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand the study and voluntarily sign the informed consent form;
2. Age between 18 and 75 years;
3. Histologically confirmed resectable or potentially resectable locally advanced gastric/gastroesophageal junction adenocarcinoma;
4. Tumor Regression Grade (TRG) 2 or 3 after preoperative adjuvant therapy;
5. R0 resection after neoadjuvant chemotherapy;
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1;
7. Life expectancy of at least 2 years;
8. No prior anti-cancer treatment received;
9. Good compliance and cooperation with follow-up.

Exclusion Criteria:

1. Inability to comply with the study protocol or procedures;
2. History of prior gastric cancer surgery;
3. Contraindications to surgical treatment and chemotherapy or physical condition and organ function that do not allow for major abdominal surgery;
4. Distant metastasis to organs other than the liver, such as lung, brain, and bone;
5. Known HER2-positive patients;
6. Uncontrolled hypertension despite medication prior to enrollment;
7. Poorly controlled diabetes despite medication prior to enrollment;
8. Urine routine indicating proteinuria ≥2+, and a 24-hour urine protein quantification >1.0g;
9. Presence of conditions requiring intervention such as bleeding, perforation, or obstruction prior to enrollment;
10. Patients deemed ineligible for this study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2023-09-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
3-year recurrence-free survival rate | Three years after surgery
  Percentage of recurrence-free patients within 3 years of surgery

SECONDARY OUTCOMES:
Overall survival | OS is the time interval from the start of treatment to death due to any reason or lost of follow-up，whichever came first, assessed up to 3 years"
  From the start of treatment to the date of death from any cause
AEs-Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | from the first drug administration to within 30 days for the last dose
  Patients' blood and non-blood abnormal values or conditions were collected according to the frequency of visits per cycle and recorded for evaluation using CTCAE5.0 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Fei Ma, M.D., Principal Investigator — Working relationship
Locations (1):
- Henan Cancer Hospital, Zhengzhou, China